CLINICAL TRIAL: NCT06870838
Title: Neuroinflammation in Frontotemporal Lobar Degeneration - a Multimodal Biomarker Study
Brief Title: Neuroinflammation in FTLD
Status: Active, not recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Matthias van Osch, Professor, Leiden University Medical Center
Other Study IDs: P21.090
Record Dates: First submitted 2025-02-03; First posted 2025-03-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-02

CONDITIONS: Corticobasal Syndrome(CBS); Primary Progressive Aphasia(PPA); Progressive Supranuclear Palsy(PSP); Behavioral Variant Frontotemporal Dementia (bvFTD); Frontotemporal Lobar Degeneration (FTLD)
Keywords: Frontotemporal lobar degeneration; Iron accumulation; 7T-MRI; Neurodegeneration; Neuroinflammation; QSM; CSF; Blood; MRS; dMRS
MeSH Terms: conditions — Corticobasal Degeneration; Aphasia, Primary Progressive; Supranuclear Palsy, Progressive; Frontotemporal Lobar Degeneration; Nerve Degeneration; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma, serum, DNA, CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patients with probable FTLD-tau: clinical diagnosis of PSP, CBS, or nfvPPA, or any clinical FTLD spectrum diagnosis with a proven MAPT mutation
  Interventions: Diagnostic Test: 7T MRI scan; Diagnostic Test: CSF; Diagnostic Test: Blood withdrawal; Diagnostic Test: Neuropsychological assessment; Diagnostic Test: Clinical measures
- Patients with probable FTLD-TDP: a clinical diagnosis of svPPA, FTLD-ALS or any clinical FTLD spectrum diagnosis with a proven GRN mutation or C9orf72 HRE
  Interventions: Diagnostic Test: 7T MRI scan; Diagnostic Test: CSF; Diagnostic Test: Blood withdrawal; Diagnostic Test: Neuropsychological assessment; Diagnostic Test: Clinical measures
- At-risk individuals: Healthy individuals with a first degree relative with a MAPT or GRN mutation or C9orf72 HRE. These subjects therefore all have a 50% risk to carry one of these genetic variants and develop FTLD later in life.
  Interventions: Diagnostic Test: 7T MRI scan; Diagnostic Test: CSF; Diagnostic Test: Blood withdrawal; Diagnostic Test: Neuropsychological assessment; Diagnostic Test: Clinical measures
- Healthy controls: Healthy individuals without increased risk to develop FTLD
  Interventions: Diagnostic Test: 7T MRI scan; Diagnostic Test: CSF; Diagnostic Test: Blood withdrawal; Diagnostic Test: Neuropsychological assessment; Diagnostic Test: Clinical measures

INTERVENTIONS:
Diagnostic Test: 7T MRI scan — MRI-scanning of the brain using a 7T MRI scanner
Diagnostic Test: CSF — CSF collection via lumbar puncture
Diagnostic Test: Blood withdrawal — Blood is collected by doing a blood withdrawal
Diagnostic Test: Neuropsychological assessment — Tests for memory, language, attention, executive functions, praxis, social cognition, visuoconstructive skills
Diagnostic Test: Clinical measures — Medical history, neurological assessment, neuropsychiatric inventory

SUMMARY:
The goal of this observational study is to investigate the role of neuroinflammation in frontotemporal lobar degeneration (FTLD). The main aims of this study are:

1. To elucidate the role and timing of neuroinflammation in FTLD by using a combination of clinical measures, 7T MRI, and CSF biomarkers;
2. To differentiate FTLD-TDP and FTLD-tau during life using biomarkers for neuroinflammation;
3. To identify biomarkers to predict and monitor disease progression in FTLD;

Secondary aim:

1. To explore the role of brain clearance in the disease process of FTLD.

Participants will undergo 7T MRI scans, blood and CSF collection, clinical, neurological, and neuropsychological evaluation.

DETAILED DESCRIPTION:
At baseline, the study will involve the following procedures: clinical assessment including neurological and neuropsychological investigation, blood sampling, and a voluntarily lumbar puncture on the first day at the Erasmus MC University Medical Center, (EMC) and two sessions of 7T MRI scanning on the second day at the Leiden University Medical Center (LUMC). After one year, clinical assessment and blood analyses will be repeated in the EMC to assess disease progression. The aim is to include 25 patients with probable or definite FTLD-tau, 25 patients with probable or definite FTLD-TDP, 50 healthy individuals with 50% risk to carry a mutation in MAPT or GRN, or the C9orf72 HRE. If necessary for age matching, 10 additional healthy subjects without increased risk of FTLD will be included.

ELIGIBILITY:
Inclusion Criteria:

* Ability to undergo MRI scanning
* For probable FTLD-tau: a clinical diagnosis of PSP, CBS or nfvPPA, or any clinical FTLD spectrum diagnosis with a proven MAPT mutation
* For probable FTLD-TDP: a clinical diagnosis of svPPA or any clinical FTLD spectrum diagnosis with a proven GRN mutation or C9orf72 repeat expansion
* For presymptomatic mutation carriers: a MAPT mutation, GRN mutation or a C9orf72 mutation without clinical sign of a FTLD spectrum phenotype (CDR 0) For control subjects: no known neurological or psychiatric disorder
* For controls: no known neurological or psychiatric disorder

Exclusion Criteria:

* Other neurological or psychiatric disorder that may affect cognitive functions, such as a brain tumour, multiple sclerosis or drug or alcohol abuse or use of psycho-active medications
* CSF profile (β-amyloid, p-tau, t-tau) suggestive of AD pathology
* Clinical dementia Rating Scale (CDR) score >1
* Contra-indication to undergo MRI
* Contra-indication to undergo lumbar puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with probable FTLD-tau (n =25) are defined as a clinical diagnosis of PSP, CBS, or nfvPPA, or any clinical FTLD spectrum diagnosis with a proven MAPT mutation. In patients with CBS or nfvPPA, CSF analyses and genetic screening will be used to rule out underlying AD pathology or having a pathogenetic variant causing FTLD-TDP pathology. Patients with probable FTLD-TDP (n=25) are indicated by either a clinical diagnosis of svPPA, FTLD-ALS or any clinical FTLD spectrum diagnosis with a proven GRN mutation or C9orf72 HRE.
  At-risk individuals (n=50) will be recruited through our ongoing FTD-RisC project. These individuals have no clinical signs of an FTLD phenotype, but have a first degree relative with genetic FTLD. These subjects have 50% risk to carry one of the genetic variants. Through anonymous genetic screening, this group will be divided into presymptomatic mutation carriers and healthy individuals. If necessary for age-matching, 10 healthy controls will be included.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
MR Spectroscopy in the lateral anterior cingulate cortex | At baseline
  MR Spectroscopy data analysis in a single volume of interest in the lateral anterior cingulate cortex to assess changes in metabolites related to neurodegeneration and neuroinflammation. The analysis in LCModel will give us metabolite concentrations for total N-acetyl-aspertate (tNAA), glutamate (Glu), myo-inositol (mI), and total choline compound (tCho).
Diffusion weighted MR spectroscopy in the lateral anterior cingulate cortex | At baseline
  Diffusion weighted MR Spectroscopy data analysis in a single volume of interest in the lateral anterior cingulate cortex to assess changes in the apparent diffusion coefficients of specific metabolites related to neurodegeneration and neuroinflammation. The analysis done in LCModel will give us metabolite apparent diffusion coefficients for total N-acetyl-aspertate (tNAA), glutamate (Glu), myo-inositol (mI), and total choline compound (tCho).
Quantitative susceptibility mapping for iron localization and quantification | At baseline
  Cross-sectional MR analysis to determine iron accumulation in the brain. The analysis will be performed with the SEPIA toolbox to obtain quantitative susceptibility values in various brain regions.
Neurodegeneration biomarkers in blood | At baseline
  Biomarkers for neurodegeneration (neurofilament light chain (NFL), total tau) in blood.
Neurodegeneration biomarkers in CSF | At baseline
  Biomarkers for neurodegeneration (neurofilament light chain (NFL), total tau) in CSF.
Neuroinflammation biomarkers in CSF | At baseline
  Biomarkers for neuroinflammation (YKL-40, TREM-1, TREM-2, IL-1, IL-6, TNF-α, GFAP, CHIT1) in CSF.
Iron accumulation biomarkers in blood | At baseline
  Biomarkers for iron accumulation ( ferritin, and iron) in blood.
Iron acccumulation biomarkers in CSF | At baseline
  Biomarkers for iron accumulation (transferritin, ferritin, and iron) in CSF.

SECONDARY OUTCOMES:
Clinical and neuropsycological evaluation: Clinical dementia rating scale | At baseline and 1 year follow-up
  Cognitive and neuropsychological assessments for clinical dementia rating scale (CDR) to assess the cognitive functioning of the participant. The CDR is a combination score including multiple neuropsychological functioning on multiple domains (memory, language, attention, executive function, praxis, social cognition, and visuoconstructive skills) and clinical evaluation. A score of 0 means not impaired or no symptoms, a score of 0.5 means prodromal, and a score of 1 and higher (up to 3) reflects a symptomatic individual.
Clinical and neuropsycological evaluation: Montreal Cognitive Assessment | At baseline and 1 year follow-up
  Cognitive and neuropsychological assessments for Montreal Cognitive Assessment (MoCA) to assess the cognitive functioning of the participant. A total score of 30 can be obtained. A higher score reflects a better performance. The cut-off point for a normal score is 26. A score lower than 26 reflects impairments or one or more cognitive domains.
Clinical evaluation: Parkinson's Disease Rating Score | At baseline and 1 year follow-up
  Neurological examination for Unified Parkinson's Disease rating score (UPDRS). The score will be between 0 and 260, with a lower score indicating no symptoms and a total score of 260 indicating all symptoms.
Clinical evaluation: Neuropsychiatric assessment | At baseline and 1 year follow-up
  Neuropsychiatric examination with the neuropsychiatric inventory (NPI) to assess psychiatric symptoms. The NPI has a total score range of [0, 144], with a higher score indicating more neuropsychiatric symptoms. A NPI score higher than 0 indicates the presence of one or more symptoms, a score of 4 or higher indicates moderate symptoms.

OTHER OUTCOMES:
7T MR markers for brain clearance: CSF mobility | At baseline
  Assessment of the CSF mobility in the perivascular spaces throughout the brain using a T2-weighted scan and diffusion weighted scans.
7T MRI markers for brain clearance: prevalance of perivascular spaces | At baseline
  In this analysis, the visible perivascular spaces on a T2-weighted scan (0.6 x 0.6 x 0.6 mm) will be counted and their volume will be calculated to assess changes in the different groups.
Markers for brain clearance: CSF | At baseline
  Levels of total tau and AQP4

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prinse FAM, van der Weerd L, van Swieten JC, Ronen I, Seelaar H, Hirschler L, Najac C, Dopper EGP. Investigating the role of neuroinflammation and brain clearance in frontotemporal lobar degeneration using 7T MRI and fluid biomarkers: protocol for a cross-sectional study in a tertiary care setting. BMJ Open. 2025 Aug 3;15(8):e102668. doi: 10.1136/bmjopen-2025-102668. PMID 40754329